CLINICAL TRIAL: NCT05874128
Title: PROSPECTIVE EVALUATION OF HEARTFOCUS: A SOFTWARE SUPPORTING THE ACQUISITION OF CARDIAC ULTRASOUND EXAMS (HF-01)
Brief Title: PROSPECTIVE EVALUATION OF HEARTFOCUS
Acronym: HF-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DESKi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HF-01
Record Dates: First submitted 2023-05-05; First posted 2023-05-24 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Disease
Keywords: Cardiac disease; Novices; Guidance; Artificial intelligence; Ejection Fraction; Ultrasound
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Study participants (Experimental): 240 patients will be included, 120 in Site 01 (Bordeaux) and 120 in Site 02 (New York)
  Interventions: Device: Using HeartFocus software with AI guidance (Novices); Device: Using HeartFocus software without AI-guidance

INTERVENTIONS:
Device: Using HeartFocus software with AI guidance (Novices) — The novice are nurses without prior ultrasound experience performed limited echocardiograms using the HeartFocus AI-based guidance software (DESKi). After a half-day training and practice on ≤9 patients, each novice acquired echocardiographic clips for 10 standard transthoracic views with the assistance of real-time software guidance and automated recording.
Device: Using HeartFocus software without AI-guidance — Experienced sonographers and cardiologists performed limited echocardiograms using HeartFocus software, without AI assistance. The experts acquired echocardiographic sequences corresponding to the 10 standard transthoracic views, just like the novices.

SUMMARY:
The study's objective is to evaluate if exams, performed with the HeartFocus software by novices, are of sufficient quality to visually analyze the left ventricular size, the left ventricular function, the right ventricular size, and the presence of non-trivial pericardial effusion.

Novices will be nurses without prior ultrasound experience who have received dedicated training on cardiac ultrasound and on Heartfocus software. Ultrasound exams will be limited to the acquisition of 10 reference views

DETAILED DESCRIPTION:
This prospective multicentric international pivotal trial will evaluate the ability of the Heartfocus software to support novices for the acquisition of 10 reference views of cardiac ultrasound. The 10 reference views are the following:

Parasternal long axis, Parasternal short axis at the aortic valve, Parasternal short axis at the mitral valve Parasternal short axis at the papillary muscles Apical 5-chamber, Apical 4-chamber, Apical 3-chamber, Apical 2-chamber, Subcostal 4-chamber, Subcostal inferior vena cava.

Patients included in the study will be adult patients scheduled for an echocardiogram at one of the two investigating centers. Ultrasound exams will be limited to the acquisition 10 reference views.

Patients will receive 2 additional limited exams, which consist of the acquisition of ultrasound clips for each of the 10 references views:

one by a novice, nurses having received a dedicated training of 2 days, with an ultrasound probe and the HeartFocus software with the guidance system, one by an expert (experienced sonographer/cardiologist) with the same ultrasound probe and the HeartFocus software without the guidance system.

A total of 8 novices will perform the acquisition on 30 patients each. In total 240 patients will be included in the study, half in each investigator center. The exams (240 acquired by novices, 240 by experts) will be analyzed by cardiologists to assess their quality. The endpoints are described below.

ELIGIBILITY:
Inclusion Criteria:

Patient (male or female) over 18 years old, Patient having an echocardiography examination scheduled in one of the two investigation centers.

Patient who has given his non-objection to participate in the research

Exclusion Criteria:

Patient subject to a measure of legal protection (safeguard of justice, guardianship or curatorship), Patient deprived of liberty by judicial or administrative decision, Patient being unable to give his non-objection, Pregnant or breastfeeding women, Patient with cardiac anatomy that does not allow reference electrocardiographic sections to be made (situs inversus, single ventricle, congenital anomalies, etc), Patient having benefited from prior echocardiographic exams whose reports mention poor or weak echogenicity, Patient having known chest deformity that has already been mentioned in previous reports or has been the subject of investigations (pectum excavatum), Patient who has undergone total or partial pneumectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biana Trost, MD, FACC, FASE, Principal Investigator — Department of Cardiology Lenox Hill Hospital
Locations (2):
- Lenox Hill Hospital, New York, New York, United States
- University Hospital of Bordeaux, Bordeaux, Aquitaine, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients (≥18 years) scheduled for a clinically indicated echocardiogram were consecutively recruited at two academic medical centers: University Hospital of Bordeaux (France) and Lenox Hill Hospital (New York, USA). Recruitment occurred between november 2023 and august 2024.
Pre-assignment Details: A total of 247 patients were screened. Of these, 246 provided informed consent; among these, 6 participants withdrew before undergoing the study echocardiography. Reasons included withdrawal of consent (n=3), scheduling conflicts (n=2), and technical difficulties (n=1). Thus, 240 patients were finally enrolled in this study, meaning that they completed both novice and expert echocardiography exams and were included in the Full Analysis Set.
Groups:
- Participants: 240 patients will be included, 120 in Site 01 (Bordeaux) and 120 in Site 02 (New York). They all received two limited exams: one administered by a novice, and the other by an expert.
Period: Overall Study
Arm/Group | Participants
Started | 240
Completed | 240
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Each participant may be presented with several prior cardiac and noncardiac diagnoses
Groups:
- France: This group consisted of 120 patients enrolled at the participating University Hospital of Bordeaux, France.
- United States: This group consisted of 120 patients enrolled at Lenox Hill Hospital, New York, United States.
- Total: Total of all reporting groups
Arm/Group | France | United States | Total
Number analyzed (Participants) | 120 | 120 | 240
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 70 | 117
  Male | 73 | 50 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 18 | 18
  Not Hispanic or Latino | 0 | 90 | 90
  Unknown or Not Reported | 120 | 12 | 132
BMI (Body Mass Index) [Count of Participants; unit: Participants]
  <25 | 56 | 41 | 97
  ≤25-30 | 44 | 49 | 93
  ≥30 | 20 | 30 | 50
Race [Count of Participants; unit: Participants]
  White | 0 | 52 | 52
  Black/African American | 0 | 36 | 36
  Asian | 0 | 3 | 3
  American Indian/Alaska Native | 0 | 0 | 0
  Unknown/not reported | 120 | 11 | 131
  Other | 0 | 18 | 18
Age, Customized [Mean (Full Range); unit: Years] | 64.7 [22 to 94] | 60.5 [22 to 87] | 62.6 [22 to 94]
Prior cardiac diagnoses [Number; unit: Percentage of participants (%)]
  Hypertension | 28.3 | 55.0 | 41.7
  Hyperlipidemia | 21.7 | 58.3 | 40.0
  Diabetes | 15.8 | 19.2 | 17.5
  Heart failure | 6.7 | 11.7 | 9.2
  Atrial fibrillation | 20.8 | 8.3 | 14.6
  Other arrhythmias | 7.5 | 7.5 | 7.5
  Coronary artery disease | 25.0 | 15.8 | 20.4
  Prior heart attack | 11.7 | 0.0 | 5.8
  Valvular heart disease | 25.8 | 9.2 | 17.5
  Pulmonary hypertension | 3.3 | 2.5 | 2.9
  Heart transplant | 3.3 | 0.8 | 2.1
  Cardiomyopathies | 15.0 | 5.8 | 10.4
  Congenital heart disease | 0.0 | 0.8 | 0.4
  Other | 4.2 | 10.0 | 7.1
  None | 17.5 | 17.5 | 17.5
  Not reported | 0.8 | 0.8 | 0.8
Prior noncardiac diagnoses [Number; unit: Percentage of participants (%)]
  Renal disease | 9.2 | 10.0 | 9.6
  COPD/emphysema | 5.0 | 4.2 | 2.9
  Pulmonary embolus | 1.7 | 4.2 | 2.9
  Systemic infiltrative disease | 0 | 0.8 | 0.4
  Cancer | 18.3 | 21.7 | 20.0
  Underwent chemotherapy | 1.7 | 10.0 | 5.8
  Underwent radiation | 2.5 | 2.5 | 2.5
  Other | 22.5 | 38.3 | 30.4
  None | 48.3 | 36.7 | 42.5
  Not reported | 0.8 | 2.5 | 1.7

OUTCOME MEASURES:

1. Primary Outcome: The Left Ventricular Size (Qualitative Visual Assessment)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the exam had sufficient image quality to allow visual analysis of left ventricular size. Each exam was independently reviewed by five cardiologists. If at least three cardiologists rated the exam as "Yes" (sufficient quality), the exam was classified as having sufficient image quality; if at least three rated it as "No", the exam was classified as not sufficient. The results represent the percentage of scans evaluated as having sufficient image quality.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: All 240 participants received two ultrasound examinations: one performed by novice operators using HeartFocus AI Guidance, and one performed by expert operators using HeartFocus without AI Guidance. Therefore, the 240 individuals included in the 'Novice' and 'Expert' result groups are the same participants. The groups were separated solely to present the performance results obtained by novices versus experts on the same 240 participants, not because they represent distinct populations.
Measure: Number (95% Confidence Interval); unit: Percentage of scans obtained (%)
Groups:
- Novice With AI Guidance: Nurses without prior ultrasound experience performed limited echocardiograms using the HeartFocus AI-based guidance software (DESKi). After a half-day training and practice on ≤9 patients, each novice acquired echocardiographic clips for 10 standard transthoracic views with the assistance of real-time software guidance and automated recording.
- Expert Without AI Guidance: Experienced sonographers or cardiologists performed limited echocardiograms using HeartFocus software without AI assistance. Experts acquired echocardiographic clips for the same 10 standard transthoracic views as the novices.
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of scans obtained (%) | 100 [98.4 to 100] | 100 [98.4 to 100]

2. Primary Outcome: The Left Ventricular Function (Qualitative Visual Assessment)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the ultrasound examination had sufficient image quality to allow visual analysis of left ventricular function. Each exam was independently reviewed by five cardiologists. If at least three cardiologists rated the exam as "Yes" (sufficient quality), the exam was classified as having sufficient image quality; if at least three rated it as "No", the exam was classified as not sufficient. The results represent the percentage of scans evaluated as having sufficient image quality.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of scans obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of scans obtained (%) | 100 [98.4 to 100] | 100 [98.4 to 100]

3. Primary Outcome: The Right Ventricle Size (Qualitative Visual Assessment)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the ultrasound examination had sufficient image quality to allow visual analysis of right ventricular size. Each exam was independently reviewed by five cardiologists. If at least three cardiologists rated the exam as "Yes" (sufficient quality), the exam was classified as having sufficient image quality; if at least three rated it as "No", the exam was classified as not sufficient. The results represent the percentage of scans evaluated as having sufficient image quality.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of scans obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of scans obtained (%) | 100 [98.4 to 100] | 100 [98.4 to 100]

4. Primary Outcome: The Presence of Non-trivial Pericardial Effusion (Qualitative Visual Assessment)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the ultrasound exam had sufficient image quality to visually analyze the presence of non-trivial pericardial effusion. Each exam was independently reviewed by five cardiologists. If at least three cardiologists rated the exam as 'Yes' (sufficient quality), the exam was classified as having sufficient image quality; if at least three rated it as 'No', the exam was classified as not sufficient. The results represent the percentage of scans evaluated as having sufficient image quality.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of scans obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of scans obtained (%) | 100 [98.4 to 100] | 100 [98.4 to 100]

5. Secondary Outcome: The Function of the Right Ventricle (Qualitative Visual Assessment)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the ultrasound examination had sufficient image quality to allow visual analysis of right ventricular function. Each exam was independently reviewed by five cardiologists. If at least three cardiologists rated the exam as 'Yes' (sufficient quality), the exam was classified as having sufficient image quality; if at least three rated it as 'No', the exam was classified as not sufficient. The results represent the percentage of scans evaluated as having sufficient image quality.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of scans obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of scans obtained (%) | 99.6 [97.7 to 99.9] | 100 [98.4 to 100]

6. Secondary Outcome: The Left Atrium Size (Qualitative Visual Assessment)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the ultrasound examination had sufficient image quality to allow visual analysis of left atrium size. Each exam was independently reviewed by five cardiologists. If at least three cardiologists rated the exam as 'Yes' (sufficient quality), the exam was classified as having sufficient image quality; if at least three rated it as 'No', the exam was classified as not sufficient. The results represent the percentage of scans evaluated as having sufficient image quality.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of scans obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of scans obtained (%) | 100 [98.4 to 100] | 100 [98.4 to 100]

7. Secondary Outcome: The Right Atrium Size (Qualitative Visual Assessment)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the ultrasound examination had sufficient image quality to allow visual analysis of right atrium size. Each exam was independently reviewed by five cardiologists. If at least three cardiologists rated the exam as 'Yes' (sufficient quality), the exam was classified as having sufficient image quality; if at least three rated it as 'No', the exam was classified as not sufficient. The results represent the percentage of scans evaluated as having sufficient image quality.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of scans obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of scans obtained (%) | 98.8 [96.4 to 99.6] | 100 [98.4 to 100]

8. Secondary Outcome: The Segmental Kinetics of the Left Ventricle (Qualitative Visual Assessment)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the ultrasound examination had sufficient image quality to allow visual analysis of the segmental kinetics of the left ventricle. Each exam was independently reviewed by five cardiologists. If at least three cardiologists rated the exam as 'Yes' (sufficient quality), the exam was classified as having sufficient image quality; if at least three rated it as 'No', the exam was classified as not sufficient. The results represent the percentage of scans evaluated as having sufficient image quality.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of scans obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of scans obtained (%) | 95.4 [92.0 to 97.4] | 100 [98.4 to 100]

9. Secondary Outcome: The Aortic Valve (Qualitative Visual Assessment)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the ultrasound examination had sufficient image quality to allow visual analysis of the aortic valve. Each exam was independently reviewed by five cardiologists. If at least three cardiologists rated the exam as 'Yes' (sufficient quality), the exam was classified as having sufficient image quality; if at least three rated it as 'No', the exam was classified as not sufficient. The results represent the percentage of scans evaluated as having sufficient image quality.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of scans obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of scans obtained (%) | 98.8 [96.4 to 99.6] | 100 [98.4 to 100]

10. Secondary Outcome: The Mitral Valve (Qualitative Visual Assessment)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the ultrasound examination had sufficient image quality to allow visual analysis of the mitral valve. Each exam was independently reviewed by five cardiologists. If at least three cardiologists rated the exam as 'Yes' (sufficient quality), the exam was classified as having sufficient image quality; if at least three rated it as 'No', the exam was classified as not sufficient. The results represent the percentage of scans evaluated as having sufficient image quality.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of scans obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of scans obtained (%) | 100 [98.4 to 100] | 100 [98.4 to 100]

11. Secondary Outcome: The Tricuspid Valve (Qualitative Visual Assessment)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the ultrasound examination had sufficient image quality to allow visual analysis of the tricuspid valve. Each exam was independently reviewed by five cardiologists. If at least three cardiologists rated the exam as 'Yes' (sufficient quality), the exam was classified as having sufficient image quality; if at least three rated it as 'No', the exam was classified as not sufficient. The results represent the percentage of scans evaluated as having sufficient image quality.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of scans obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of scans obtained (%) | 95.4 [92.0 to 97.4] | 99.2 [97.0 to 99.8]

12. Secondary Outcome: The Size of Inferior Vena Cava (Qualitative Visual Assessment)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the ultrasound examination had sufficient image quality to allow visual analysis of the size of the inferior vena cava. Each exam was independently reviewed by five cardiologists. If at least three cardiologists rated the exam as 'Yes' (sufficient quality), the exam was classified as having sufficient image quality; if at least three rated it as 'No', the exam was classified as not sufficient. The results represent the percentage of scans evaluated as having sufficient image quality.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of scans obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of scans obtained (%) | 78.3 [72.7 to 83.1] | 98.3 [95.8 to 99.4]

13. Secondary Outcome: Apical-2-Chamber (Diagnostic Quality Clip)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the Apical-2-Chamber (A2C) clip had sufficient image quality for interpretation, in order to determine the entire endocardial contour of the left ventricle, calculate ejection fraction by Simpson's method, and detect wall motion abnormalities. Each clip was independently reviewed by five cardiologists. If at least three cardiologists rated the clip as 'Yes' (sufficient quality), the clip was classified as a Diagnostic Quality Clip (DQC); if at least three rated it as 'No', the clip was classified as not sufficient. The results represent the percentage of Diagnostic Quality Clips (DQC) obtained.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of DQC obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of DQC obtained (%) | 82.5 [77.2 to 86.8] | 98.3 [95.8 to 99.4]

14. Secondary Outcome: Apical-3-Chamber (Diagnostic Quality Clip)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the Apical-3-Chamber (A3C) clip had sufficient image quality for interpretation, in order to determine the endocardial definition of the left ventricle, detect wall motion abnormalities, and ensure that the right ventricle and aortic valve leaflets were correctly visualized. Each clip was independently reviewed by five cardiologists. If at least three cardiologists rated the clip as 'Yes' (sufficient quality), the clip was classified as a Diagnostic Quality Clip (DQC); if at least three rated it as 'No', the clip was classified as not sufficient. The results represent the percentage of Diagnostic Quality Clips (DQC) obtained.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of DQC obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of DQC obtained (%) | 90 [85.6 to 93.2] | 100 [98.4 to 100]

15. Secondary Outcome: Apical-4-Chamber (Diagnostic Quality Clip)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the Apical-4-Chamber (A4C) clip had sufficient image quality for interpretation, in order to determine the entire endocardial contour of the left ventricle, calculate ejection fraction by Simpson's method, and detect wall motion abnormalities. Each clip was independently reviewed by five cardiologists. If at least three cardiologists rated the clip as 'Yes' (sufficient quality), the clip was classified as a Diagnostic Quality Clip (DQC); if at least three rated it as 'No', the clip was classified as not sufficient. The results represent the percentage of Diagnostic Quality Clips (DQC) obtained.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of DQC obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of DQC obtained (%) | 96.2 [93.0 to 98.0] | 100 [98.4 to 100]

16. Secondary Outcome: Apical-5-Chamber (Diagnostic Quality Clip)
Description: "For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the Apical-5-Chamber (A5C) clip had sufficient image quality for interpretation, in order to determine the endocardial definition of the left ventricle and ensure proper visualization of the outflow chamber and aortic valve. Each clip was independently reviewed by five cardiologists. If at least three cardiologists rated the clip as 'Yes' (sufficient quality), the clip was classified as a Diagnostic Quality Clip (DQC); if at least three rated it as 'No', the clip was classified as not sufficient. The results represent the percentage of Diagnostic Quality Clips (DQC) obtained.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of DQC obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of DQC obtained (%) | 93.3 [89.4 to 95.9] | 99.2 [97.0 to 99.8]

17. Secondary Outcome: Parasternal Long Axis (Diagnostic Quality Clip)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the Parasternal Long-Axis (PLAX) clip had sufficient image quality for interpretation, in order to ensure that the basal segments of the left ventricle were visible with adequate image quality for diameter measurement and detection of wall motion abnormalities, and to confirm that the long axis, aortic valve, and right ventricle were correctly visualized to consider the view as a good PLAX. Each clip was independently reviewed by five cardiologists. If at least three cardiologists rated the clip as 'Yes' (sufficient quality), the clip was classified as a Diagnostic Quality Clip (DQC); if at least three rated it as 'No', the clip was classified as not sufficient. The results represent the percentage of Diagnostic Quality Clips (DQC) obtained.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of DQC obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of DQC obtained (%) | 97.5 [94.7 to 98.8] | 100 [98.4 to 100]

18. Secondary Outcome: Parasternal Short Axis Aortic (Diagnostic Quality Clip)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the Parasternal Short-Axis Aortic (PSAX-AV) clip had sufficient image quality for interpretation, in order to ensure adequate image quality to visualize the aortic valve leaflets. Each clip was independently reviewed by five cardiologists. If at least three cardiologists rated the clip as 'Yes' (sufficient quality), the clip was classified as a Diagnostic Quality Clip (DQC); if at least three rated it as 'No', the clip was classified as not sufficient. The results represent the percentage of Diagnostic Quality Clips (DQC) obtained.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of DQC obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of DQC obtained (%) | 89.2 [84.6 to 92.5] | 99.2 [97.0 to 99.8]

19. Secondary Outcome: Parasternal Short Axis Mitral (Diagnostic Quality Clip)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the Parasternal Short-Axis Mitral (PSAX-MV) clip had sufficient image quality for interpretation, in order to ensure adequate image quality to detect wall motion abnormalities and visualize valvular movement. Each clip was independently reviewed by five cardiologists. If at least three cardiologists rated the clip as 'Yes' (sufficient quality), the clip was classified as a Diagnostic Quality Clip (DQC); if at least three rated it as 'No', the clip was classified as not sufficient. The results represent the percentage of Diagnostic Quality Clips (DQC) obtained.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of DQC obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of DQC obtained (%) | 90.8 [86.5 to 93.9] | 99.6 [97.7 to 99.9]

20. Secondary Outcome: Parasternal Short Axis Papillary Muscles (Diagnostic Quality Clip)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the Parasternal Short-Axis Papillary Muscles (PSAX-PM) clip had sufficient image quality for interpretation, in order to ensure adequate image quality to detect wall motion abnormalities, visualize valvular movement, and visualize both papillary muscles. Each clip was independently reviewed by five cardiologists. If at least three cardiologists rated the clip as 'Yes' (sufficient quality), the clip was classified as a Diagnostic Quality Clip (DQC); if at least three rated it as 'No', the clip was classified as not sufficient. The results represent the percentage of Diagnostic Quality Clips (DQC) obtained.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of DQC obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of DQC obtained (%) | 97.1 [94.1 to 98.6] | 99.2 [97.0 to 99.8]

21. Secondary Outcome: Sub Costal-4-Chamber (Diagnostic Quality Clip)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the Subcostal 4-Chamber (SC-4C) clip had sufficient image quality for interpretation, in order to ensure adequate image quality for detecting a pericardial effusion between the right ventricle and liver. Full visualization of the left and right ventricles was not required. Each clip was independently reviewed by five cardiologists. If at least three cardiologists rated the clip as 'Yes' (sufficient quality), the clip was classified as a Diagnostic Quality Clip (DQC); if at least three rated it as 'No', the clip was classified as not sufficient. The results represent the percentage of Diagnostic Quality Clips (DQC) obtained.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of DQC obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of DQC obtained (%) | 89.2 [84.6 to 92.5] | 98.3 [95.8 to 99.4]

22. Secondary Outcome: Sub Costal Inferior Vena Cava (Diagnostic Quality Clip)
Description: For each participant, one novice and one expert performed a limited echocardiographic exam on the same patient, so that the quality of each exam could be evaluated by cardiologists. Blinded cardiologists evaluated whether the Subcostal Inferior Vena Cava (SC-IVC) clip had sufficient image quality for interpretation, in order to ensure adequate image quality to measure the diameter of the IVC a few centimeters before it reaches the heart. Each clip was independently reviewed by five cardiologists. If at least three cardiologists rated the clip as 'Yes' (sufficient quality), the clip was classified as a Diagnostic Quality Clip (DQC); if at least three rated it as 'No', the clip was classified as not sufficient. The results represent the percentage of Diagnostic Quality Clips (DQC) obtained.
Time Frame: Images evaluated by the cardiologists after the acquisition
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of DQC obtained (%)
Arm/Group | Novice With AI Guidance | Expert Without AI Guidance
Number analyzed (Participants) | 240 | 240
Percentage of DQC obtained (%) | 77.5 [71.8 to 82.3] | 98.3 [95.8 to 99.4]

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, approximately up to one hour
Description: Adverse events, adverse reactions, device deficiencies, and incidents must be reported to the different health vigilance circuits applicable to each product or practice concerned in accordance with the regulations in force. In addition, three standardized reporting forms have been implemented for this study: one for adverse events (AE), one for serious adverse events (SAE), and one for device deficiencies. These forms ensure consistent data collection and facilitate timely reporting and analysis
Arm/Group | Participants
All-Cause Mortality (participants affected / at risk) | 0/240
Serious Adverse Events (participants affected / at risk) | 0/240
Other Adverse Events (participants affected / at risk) | 0/240

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-12-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT05874128/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT05874128/SAP_001.pdf